CLINICAL TRIAL: NCT05717231
Title: The Effect of Laughter Yoga on Tex Anxiety and Educational Stress in 8th-Grade Students
Brief Title: The Effect of Laughter Yoga on Tex Anxiety and Educational Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Bilge Kalanlar, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: E2273
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Laughter Therapy; Anxiety; Stress, Exam
MeSH Terms: conditions — Anxiety Disorders | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laughter yoga (Experimental): Laughter yoga was performed face-to-face with the intervention group for 35-40 minutes twice a week and in 6 sessions in total.
  Interventions: Behavioral: laughter yoga
- Control group (No Intervention): No intervention was performed for the control group

INTERVENTIONS:
Behavioral: laughter yoga — laughter yoga
  Arms: laughter yoga

SUMMARY:
The primary purpose of this study is to examine the effects of laughter therapy on tex anxiety and educational stress in 8th-grade students.

ELIGIBILITY:
The inclusion criteria of the study were determined as being an 8th-grade student, speaking and understanding Turkish, and being able to perform daily life activities.

The exclusion criteria of the study were to have undergone a surgical operation in the last three months, and to have uncontrollable blood pressure, diabetes and asthma.

Ages: 13 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2022-04-03 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Westside Test Anxiety Scale | up to 6 weeks
  The Westside Test Anxiety Inventory is a ten-item scale in a single dimension that aims to measure test anxiety. The scale was developed to be used in examining the effect of a program to reduce test anxiety.

SECONDARY OUTCOMES:
Educational stress | up to 6 weeks
  It is a self-reported 5-point Likert-type measurement tool consisting of 16 items. The educational stress scale consists of four sub-dimensions: work pressure, course load, success anxiety, and expectation versus hopelessness. In addition to the sub-dimensions in the scale, the total score for the overall scale is calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Bilge KALANLAR, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No